CLINICAL TRIAL: NCT06765174
Title: Drain Vs No Drain After Thyroid Surgeries: a Prospective Randomized Clinical Trial.
Brief Title: Randomized Controlled Trial Comparing Drains Usage Vs Without Drains After Thyroid Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Helmy Khaled Helmy, Helmy khaled helmy, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Drains Post thyroidectomy
Record Dates: First submitted 2024-12-24; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Surgery; Drains; Post Thyroidectomy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group drain (A) (Active Comparator): Drain placement post thyroid surgery
  Interventions: Device: Suction Drain placement (Example: Q-vac)
- Group no drain (B) (No Intervention): No drain placement post thyroid surgery

INTERVENTIONS:
Device: Suction Drain placement (Example: Q-vac) — After thyroid surgery we pust drain at bed of surgery to monitor post operative bleeding.
  Arms: Group drain (A)

SUMMARY:
The aim of this study is to compare patients who used drain to patients who did not use drain post-thyroidectomy regarding the short-term outcomes .

ELIGIBILITY:
Inclusion Criteria:

* (1) Male or female patients undergoing thyroidectomy (2) Patients with ages: from 18 to 60 years old. (3) Patients with normal thyroid function tests (4) Patients who are fit for general-anesthesia.

Exclusion Criteria:

* (1) Patients with bleeding diathesis and those on anticoagulants. (2) Patients with thyrotoxicosis (uncontrolled) (3) Patients those requiring neck L.N dissection. (4) Patients with previous neck surgeries. (5) Patients with severe comorbid conditions with high risk for general anesthesia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Rate of hematoma post-operative . | 24 hours
  Rate of post operative hematoma formation and effect of drain in preventing it

SECONDARY OUTCOMES:
Rate of infection | 7 days
  Compare Rate of surgical site infection between two groups
Rate of re intervention | 7 days
Post-operative pain by visual analogue scale | 3 days
Post-operative hospital stay in days | 7 days
  Length of hospital stay: described as the length of a single hospitalization, which is determined by subtracting the day of admission from the day of discharge. Data are collected from patients underwent thyroid surgery using a pretested, structured interviewer-administered questionnaire, medical record review,
Patient satisfaction by likert scale | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Abdel ghafour, Study Director — Affiliated

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Materazzi G, Ambrosini CE, Fregoli L, De Napoli L, Frustaci G, Matteucci V, Papini P, Bakkar S, Miccoli P. Prevention and management of bleeding in thyroid surgery. Gland Surg. 2017 Oct;6(5):510-515. doi: 10.21037/gs.2017.06.14. PMID 29142842
- [Background] George NM, Chitrambalam TG, Christopher PJ, Marlecha M, Selvamuthukumaran S. To drain or not to drain following thyroidectomy.: A prospective, randomized study. Saudi Med J. 2023 May;44(5):518-521. doi: 10.15537/smj.2023.44.5.20220031. PMID 37182919
- [Background] Liu J, Sun W, Dong W, Wang Z, Zhang P, Zhang T, Zhang H. Risk factors for post-thyroidectomy haemorrhage: a meta-analysis. Eur J Endocrinol. 2017 May;176(5):591-602. doi: 10.1530/EJE-16-0757. Epub 2017 Feb 8. PMID 28179452
- [Background] de Carvalho AY, Gomes CC, Chulam TC, Vartanian JG, Carvalho GB, Lira RB, Kohler HF, Kowalski LP. Risk Factors and Outcomes of Postoperative Neck Hematomas: An Analysis of 5,900 Thyroidectomies Performed at a Cancer Center. Int Arch Otorhinolaryngol. 2021 Jul;25(3):e421-e427. doi: 10.1055/s-0040-1714129. Epub 2020 Sep 30. PMID 34377179
- [Background] Musa AA, Agboola OJ, Banjo AA, Oyegunle O. The use of drains in thyroid surgery. Niger Postgrad Med J. 2010 Mar;17(1):15-8. PMID 20348976
- [Background] Portinari M, Carcoforo P. The application of drains in thyroid surgery. Gland Surg. 2017 Oct;6(5):563-573. doi: 10.21037/gs.2017.07.04. PMID 29142849
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967